CLINICAL TRIAL: NCT04116424
Title: VIGIP-SEP2: Evaluation of the Impact of the Training of Patients by a Nurse on the Adverse Drug Reaction Reporting by RRMS Patient Via a Mobile Application: Randomized Real-life Study
Acronym: VIGIP-SEP2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-022
Record Dates: First submitted 2019-10-03; First posted 2019-10-04 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-09

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nurse training of the patient (Experimental)
  Interventions: Other: nurse training of the patient
- simple information of the patient by neurologist (Active Comparator)
  Interventions: Other: neurologist accompaniement

INTERVENTIONS:
Other: nurse training of the patient — visit + telephone follow-up
  Arms: nurse training of the patient
Other: neurologist accompaniement — presentation during consultation by neurologist
  Arms: simple information of the patient by neurologist

SUMMARY:
The patient's reporting of adverse drug reactions (ADRs) is recognized as being of interest for post-marketing safety monitoring, but is still underdeveloped in France, with an average lower than the European average. A multidisciplinary team of the University Hospital of Caen, composed of neurologists and pharmacovigilants, has been carrying out since autumn 2017 a national study (VIGIP-SEP1) with 24 research centers in France (12 universitary hospitals, 6 general hospitals, and 6 private-practice neurologists) whose main objective was to evaluate the impact of multiple sclerosis (MS) patients' use of a mobile application (App) to report their ADRs. My eReport France® has been developed by the eVedrug company: ADR reports are sent by patients directly to the Regional Pharmacovigilance Centers, after analyze, clinical pharmacologist send it to the National Competent Authority. As part of VIGIP-SEP1, the accompaniment for the use of the App was carried out very simply by neurologists.

We designed a randomized controlled trial based on the assumption that a nurse training of the patient, after the initial prescription of an oral MS drug, with a telephone follow-up within 6 months, will increase by 3 times the number of patients who report ADRs compared to a simple information presented by the neurologist. The number of subjects required is 23 subjects per group.

ELIGIBILITY:
Inclusion Criteria:

* more than 18 years
* multiple sclerosis in initiation with a DMT
* patient informed and who gave informed consent

Exclusion Criteria:

* patient without mobile or tablet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
number of patients who reported at least one ADR | 3 months